CLINICAL TRIAL: NCT04754009
Title: The Effects of Trauma-sensitive Yoga and Tai Chi on Mental Health
Acronym: TSY/TC
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Northern Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-0169
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Mental Health Wellness 1
Keywords: Trauma; Depression; Anxiety; Stress; Resilience; Social Support; Alcohol consumption
MeSH Terms: conditions — Wounds and Injuries; Depression; Anxiety Disorders; Alcohol Drinking | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as Usual (TAU) (Active Comparator): Participants assigned to treatment as usual group are required to see a mental health professional for the 12 week treatment period. How often they seek counseling is up to the participant.
  Interventions: Behavioral: Treatment as Usual
- Trauma-Sensitive Yoga + TAU (Experimental): Participants assigned to the Trauma-Sensitive Yoga group will attend a 1-hour long session of yoga once a week for 12 weeks. Participants will be required to concurrently see a mental health professional for the 12 week treatment period. How often they seek counseling is up to the participant.
  Interventions: Behavioral: Trauma-Sensitive Yoga + TAU
- Chen Style Tai Chi + TAU (Experimental): Participants assigned to the Chen Style Tai Chi group will attend a 1-hour long session of tai chi once a week for 12 weeks. Participants will be required to concurrently see a mental health professional for the 12 week treatment period. How often they seek counseling is up to the participant.
  Interventions: Behavioral: Chen Style Tai Chi + TAU

INTERVENTIONS:
Behavioral: Trauma-Sensitive Yoga + TAU — Trauma-Sensitive Yoga is a movement-based approach that are used to integrate both mind and body, and promote body awareness and acceptance for those who have been exposed to traumatic events and currently experience trauma symptoms.
  Arms: Trauma-Sensitive Yoga + TAU
Behavioral: Chen Style Tai Chi + TAU — Chen Style Practical Method tai chi is a martial art that is used as a form of self-defense and to maintain physical health and well-being.
  Arms: Chen Style Tai Chi + TAU
Behavioral: Treatment as Usual — Consists of traditional talk therapy for mental health.
  Arms: Treatment as Usual (TAU)

SUMMARY:
A three-arm randomized control trial design was used to test the effectiveness of (1) Chen Style Tai Chi (TC) and talk therapy; (2) Trauma-Sensitive Yoga and talk therapy in comparison to (3) talk therapy only (control group) on four self-reported mental health outcomes: overall mental health, depression, anxiety, and trauma symptoms. Secondary outcomes include self-reported measures of resilience, stress, social support, and alcohol consumption. The two research questions driving this research study are as follows:

1. Does TSY and talk therapy significantly lower a) PTSD symptoms and b) comorbid symptoms of anxiety, depression, and other mental health determinants compared to talk therapy alone?
2. Does TC and talk therapy significantly lower a) PTSD symptoms and b) comorbid symptoms of anxiety, depression, and other mental health determinants compared to talk therapy alone?

DETAILED DESCRIPTION:
Design: This study consists of a three-arm randomized control trial design to test the effectiveness of (1) Chen Style tai chi (TC) and talk therapy; (2) trauma-sensitive yoga (TSY) and talk therapy in comparison to (3) treatment as usual (TAU), which typically consists of talk therapy, on four primary self-reported mental health outcomes: overall mental health, depression, anxiety, and trauma symptoms. Secondary outcomes include self-reported measures of resilience, stress, social support, and alcohol consumption. Other demographic information will also be collected such as race, ethnicity, education, income, family status, etc. Data collection will consist of three online assessments: a pre-test, post-test, and 1-month follow-up. In-person interviews will also be available for participants who choose to discuss their experiences.

Recruitment and Sample: Participation in these groups requires the following: 1) female gender, 2) age 18 years or older, 3) currently experiencing the symptoms of trauma, 4) an insurance carrier who can cover both individual and group mental health sessions (most in-state plans can do this), 5) paying any co-pays or deductibles associated with individual or group sessions, and 6) reliable transportation to and from appointments and group sessions.

Recruiting will take place spring 2018 to Spring 2021. Recruitment approaches include flyers, social media (e.g., Facebook), and use of MercyOne email list-serve. Those who are interested in the study will be asked to either click or enter a web link that will bring them to an online screening tool that will screen for trauma symptoms using the PTSD Checklist PCL-2 along with other questions to determine eligibility (i.e., exclusion criteria). If the participant 1) screens positive for a history of trauma according the PCL-2, answers "yes" to questions related to inclusion criteria, and answers no to questions related to the exclusion criteria, then they will be sent to a screen where they can read the full consent form. At the bottom of the page, there will be a button that allows them to choose how they want to participate in the study: 1) decline to enroll, 2) they are interested but would like to speak to a member of the research team, 3) they would like to officially enroll in the study.

Group Assignment: Participants who consent to be enrolled in the study will be randomly assigned to one of the following: (1) TSY; (2) TC or (3) TAU. Both the TSY and TC group classes will be held at the Wellness Center at the MercyOne Cedar Falls Medical Center in Cedar Falls, Iowa. Each group will meet once a week for 12 weeks for 1-hour sessions.

Assessment: If assigned to either the TC or TSY groups, we will supply participants a schedule that has the dates, times, and locations of the groups. All participants (including those in the TAU group) will then be sent a web-link to an online pre-test assessment, which should take about 20-30 minutes to complete. Participants will then attend the TC or TSY once a week for a period of 12 weeks. Those who are randomly assigned to the TAU group will be asked to see consistently see a mental health provider for the 12-week study duration. It is not specified or dictated how often participants meet with their provider nor what type of therapeutic interventions are to be used.

At the end of the 12-week study duration, all participants will be sent an online post-test assessment, with the same measures found in the pre-test. The same assessment will then be provided again in 1-month to assess for diminished effects. Participants have the option to participate in interviews where they will be asked questions about their experiences participating in the therapy group and the research study. The interviews will be audio recorded and take about 30-40 minutes to complete. These interviews are optional, and not required to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

•Women 18 years or older with a history of traumatic exposure based on the PTSD Checklist for DSM-5 screening instrument.

Exclusion Criteria

Those who:

* Find themselves frequently having uncontrolled suicidal thoughts.
* Are currently experiencing uncontrolled hallucinations or delusional thinking.
* Are cognitively unable to follow directions.
* Who have a history of sexually abusing others.
* Who have a current diagnosis of Borderline Personality Disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation of gender identify
Enrollment: 60 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Baseline in Symptoms on the Trauma Symptoms Checklist at Week 12 and 16. | Baseline and Weeks 12 and 16
  The Trauma Symptom Checklist is a validated, self-reported instrument assessing the frequency of a variety of trauma and trauma-related symptoms in the last month. Subscales include anxiety, depression, dissociation, sexual abuse trauma index, sexual problems, and sleep disturbances. Possible scores range from 0 (never occurring) to 3 (often occurring). Change = (Week 12 and 16 score - Baseline Score).
Change in Baseline in health and mental health ratings on the Medical Outcomes Study Questionnaire Short Form 36 Survey at Week 12 and 16. | Baseline and Weeks 12 and 16
  Questionnaire Short Form 36 Survey is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients. The Questionnaire Short Form 36 Survey has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0-100. Lower scores = more disability, higher scores = less disability. Change = (Week 12 and 16 score - Baseline Score).

SECONDARY OUTCOMES:
Change in Baseline Alcohol Consumption on the Alcohol Use Disorders Identification Test (AUDIT questionnaire at week 12 and 16 | Baseline and Weeks 12 and 16
  The Alcohol Consumption on the Alcohol Use Disorders Identification Test questionnaire is designed to help in the self assessment of alcohol consumption and to point out any implications for the person's health and wellbeing now and in the future. Scores for each question range from 0 to 4, with the first response for each question (e.g., never) scoring 0, the second (e.g., less than monthly) scoring 1, the third (e.g., monthly) scoring 2, the fourth (e.g., weekly) scoring 3, and the last response (eg. daily or almost daily) scoring 4. For questions 9 and 10, which only have three responses, the scoring is 0, 2 and 4 (from left to right). Lower scores = less alcohol consumption, higher scores = higher alcohol consumption. Change = (Week 12 and 16 score - Baseline Score).
Change in Baseline Resilience self-evaluation on the Brief Resilience Scale at week 12 and 16 | Baseline and Weeks 12 and 16
  The Brief Resilience Scale assesses the ability to bounce back or recover from stress. The scale consists of 6 questions, with questions 1, 3, and 5 that range from 1 (strongly disagree) to 5 (strongly agree). Questions 2, 4, 6 are rated inversely. Scoring includes adding the responses varying from 1-5 for all six items giving a range from 6-30. Divide the total sum by the total number of questions answered. Lower scores = less perceived resiliency, higher scores = higher perceived resiliency. Change = (Week 12 and 16 score - Baseline Score).
Change in Baseline Stress on the Perceived Stress Scale at week 12 and 16 | Baseline and Weeks 12 and 16
  The Perceived Stress Scale is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Lower scores = less perceived stress, higher scores = higher perceived stress. Change = (Week 12 and 16 score - Baseline Score).
Change in Baseline Pessimism/Optimism on the Life Orientation Test at week 12 and 16 | Baseline and Weeks 12 and 16
  The Life Orientation Test is a 10-item scale that measures how optimistic or pessimistic people feel about the future. Of the 10 items, 3 items measure optimism, 3 items measure pessimism, and 4 items serve as fillers. Respondents rate each item on a 4-point scale: 0 = strongly disagree, 1 = disagree, 2 = neutral, 3 = agree, and 4 = strongly agree. Lower scores = more pessimistic, higher scores = more optimistic Change = (Week 12 and 16 score - Baseline Score).
Change in Baseline on the perceived socials support Multidimensional Scale of Perceived Social Support at week 12 and 16 | Baseline and Weeks 12 and 16
  The Multidimensional Scale of Perceived Social Support is a brief research tool designed to measure perceptions of support from 3 sources: Family, Friends, and a Significant Other. The scale is comprised of a total of 12 items, with 4 items for each subscale. Respondents rate each item from a 1-7 scale, with lower scores = less perceived social support, higher scores = more perceived social support. Change = (Week 12 and 16 score - Baseline Score).

CONTACTS AND LOCATIONS:
Locations (1):
- MercyOne Cedar Falls Medical Center, Cedar Falls, Iowa, United States

IPD SHARING:
Plan to Share IPD: No